CLINICAL TRIAL: NCT04212858
Title: Amplification of Zinc- Finger Protein 217 Gene in Multiple Myeloma Patients as a Prognostic Marker
Brief Title: Amplification of Zinc Finger Protein 217 Gene in Multiple Myeloma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aya Mohammed ebrahim tawfik, specialist of clinical pathology, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: Zinc finger protein 217 gene
Record Dates: First submitted 2019-12-23; First posted 2019-12-30 (Actual); Last update posted 2019-12-30 (Actual); Status verified 2019-12

CONDITIONS: Multiple Myeloma
Keywords: Zinc finger 217 protein gene .; Multiple myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — ZNF217 protein, human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- case (Experimental): myeloma patients
  Interventions: Genetic: zinc-finger protein 217 gene
- control (Experimental): healthy control
  Interventions: Genetic: zinc-finger protein 217 gene

INTERVENTIONS:
Genetic: zinc-finger protein 217 gene — search for zinc-finger protein 217 gene in myeloma patients

SUMMARY:
Multiple myeloma (MM) is blood disorder characterized by the detection of a monoclonal paraprotein in serum or urine, which is often associated with the presence of clonal plasma cells (PCs) mainly in the bone marrow (BM) .The zinc-finger protein 217 (ZNF217) is an oncogenic protein that plays deleterious functions in various human cancers. The ZNF217 gene is located at the 20q13 chromosomal region, which is frequently amplified in human tumors .

DETAILED DESCRIPTION:
Multiple myeloma (MM) is blood disorder characterized by the detection of a monoclonal paraprotein in serum or urine, which is often associated with the presence of clonal plasma cells (PCs) mainly in the bone marrow (BM) . MM is the second most common hematologic malignancy and is expected to cause ∼13 000 new cases and 30 000 deaths in 2018. Myeloma is a genetically complex disorder characterized by multiple genetic changes, affecting different pathways, that have the ability to deregulate plasma cell biology leading to a broadly similar phenotypic manifestation of disease. From a genetic perspective, myeloma can be divided into those with and without a hyperdiploid karyotype .The zinc-finger protein 217 (ZNF217) is an oncogenic protein that plays deleterious functions in various human cancers. The ZNF217 gene is located at the 20q13 chromosomal region, which is frequently amplified in human tumors . This region also contains several oncogenes thought to confer selective advantages to cancer cells. Increased copy numbers of ZNF217 have been reported in various tumors and linked to poor outcome in some studies . ZNF217 can attenuate apoptotic signals resulting from telomere dysfunction and may promote neoplastic transformation and later stages of malignancy. ZNF217 was shown to be a prognostic biomarker and therapeutic target during breast cancer progression. In our best knowledge, No studies were done to detect ZNF217 in multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed multiple myeloma patients, who fulfill the WHO criteria of myeloma diagnosis.

Exclusion Criteria:

* Patients with any other type of malignant or benign tumors should be excluded from our study.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-02-01 (Estimated)

PRIMARY OUTCOMES:
zinc-finger protein gene 217 in myeloma patients | 2 years
  Measurement of amplification of Zinc-finger protein 217 gene in Multiple myeloma patients as a prognostic marker by fluorescence in situ hybridization technique

IPD SHARING:
Plan to Share IPD: No